CLINICAL TRIAL: NCT02747680
Title: Cerebral Responses to Insulin Induced Hypoglycemia
Acronym: 1018
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 8597
Record Dates: First submitted 2016-04-11; First posted 2016-04-22 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Type 1 Diabetes; Healthy; Hypoglycemia Unawareness
Keywords: type 1 diabetes; hypoglycemia unawareness; healthy control
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- type 1 diabetes (Other): type 1 diabetes >5 years duration Well controlled (a1c <7.5%)
  Interventions: Other: hypoglycemia (low blood sugar) in MRI
- healthy controls (Other): healthy controls
  Interventions: Other: hypoglycemia (low blood sugar) in MRI

INTERVENTIONS:
Other: hypoglycemia (low blood sugar) in MRI — hypoglycemia (low blood sugar) in MRI

SUMMARY:
This research study is designed to investigate the effect of hypoglycemia (low blood sugar) on blood flow to and biochemistry in the brain.

DETAILED DESCRIPTION:
The purpose of this study is to better understand the effect of low blood sugar (hypoglycemia) on blood flow and biochemistry in the brain. Hypoglycemia is a serious complication of diabetes treatments. It has been previously observed that hypoglycemia causes an increase in blood flow to certain parts of the brain, but it has been difficult to determine which parts of the brain specifically have an increase in blood flow. With new technology, it is now possible to determine the rate of blood flow in very small parts of the brain. The investigator expects that people with type 1 diabetes and hypoglycemia unawareness, poorly controlled diabetes, and normal subjects will have different rates of blood flow to different parts of the brain in response to hypoglycemia. Having a greater understanding of how the brain adapts to hypoglycemia may help us develop better ways to treat diabetes more safely.

ELIGIBILITY:
Inclusion Criteria:

* well controlled type 1 diabetes (hemoglobin A1C <7.5%)
* healthy controls

Exclusion Criteria:

* History of stroke, seizures, neurosurgical procedures, or arrhythmias
* Use of drugs that can alter GABA (gamma-aminobutyric acid) metabolism (such as benzodiazepines).
* Subjects must also meet requirements for a study in the magnet, which includes weight less than 300 lbs and the absence of metallic substances in their body.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2004-01 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Brain activation during euglycemia (normal blood sugar) using functional MRI | baseline
  Brain activation during euglycemia (normal blood sugar) using functional MRI
Brain activation during hypoglycemia (low blood sugar) using functional MRI | baseline
  Brain activation during hypoglycemia (low blood sugar) using functional MRI

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Seaquist, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No